CLINICAL TRIAL: NCT01507974
Title: The Efficacy of Preventive Antibiotic Treatment During the Puerperium Among Pregnant Women With Recurrent Urinary Tract Infections
Brief Title: Examination of the Efficacy of Preventive Antibiotic Treatment During the Puerperium Among Pregnant Women With Recurrent Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0068-11-EMC
Record Dates: First submitted 2012-01-04; First posted 2012-01-11 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy Complications
Keywords: preventive; antibiotic treatment; urinary tract infection; pregnancy; puerperium
MeSH Terms: conditions — Pregnancy Complications; Urinary Tract Infections | interventions — Clavulanic Acid; Trimethoprim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control arm (No Intervention): The women in this arm will not receive preventive antibiotic treatment after delivery
- preventive antibiotic treatment (Active Comparator): The women in this arm will receive preventive antibiotic treatment after the delivery to 6 weeks
  Interventions: Drug: Preventive antibiotic treatment- NITROFURANTOIN; Drug: Preventive antibiotic treatment- CEPHALEXIN; Drug: PREVENTIVE TREATMENT- AMOXICILLIN; Drug: PREVENTIVE TREATMENT- AMOXICILLIN AND CLAVULANATE POTASSIUM; Drug: PREVENTIVE TREATMENT- CEFUROXIME; Drug: PREVENTIVE TREATMENT SULFAMETHOXAZOLE AND TRIMETHOPRIM

INTERVENTIONS:
Drug: Preventive antibiotic treatment- NITROFURANTOIN — P.O NITROFURANTOIN 100 mg per day for 6 weeks
  Arms: preventive antibiotic treatment
Drug: Preventive antibiotic treatment- CEPHALEXIN — P.O CEPHALEXIN 500 MG PER DAY FOR 6 WEEKS
  Arms: preventive antibiotic treatment
Drug: PREVENTIVE TREATMENT- AMOXICILLIN — P.O AMOXICILLIN 250 MG PER DAY FOR 6 WEEKS
  Arms: preventive antibiotic treatment
Drug: PREVENTIVE TREATMENT- AMOXICILLIN AND CLAVULANATE POTASSIUM — P.O AMOXICILLIN AND CLAVULANATE POTASSIUM, 875 MG PER DAY FOR 6 WEEKS
  Arms: preventive antibiotic treatment
Drug: PREVENTIVE TREATMENT- CEFUROXIME — P.O CEFUROXIME 250 MG PER DAY FOR 6 WEEKS
  Arms: preventive antibiotic treatment
Drug: PREVENTIVE TREATMENT SULFAMETHOXAZOLE AND TRIMETHOPRIM — P.O SULFAMETHOXAZOLE AND TRIMETHOPRIM 1 TAB PER DAY FOR 6 WEEKS
  Arms: preventive antibiotic treatment

SUMMARY:
Urinary tract infection is the most common bacterial infection during pregnancy. Asymptomatic bacteriuria is the most common infection, in up to 8% of the population. Symptomatic infection may cause cystitis or cause pyelonephritis.

Among pregnant women with recurrent bacteriuria, preventive antibiotic treatment has been found to be efficacious in reducing the bacteriuria rate and the complications.

the changes of the urinary tract which appear during pregnancy usually resolve up to 3 months post-partum.

The purpose of this study is to examine the efficacy of preventive antibiotic treatment during the puerperium.

DETAILED DESCRIPTION:
During pregnancy functional modifications in the urinary tract influence the function of the urinary tract system. Those changes raise the risk of urinary tract infections. The most common bacterial infections during pregnancy are urinary tract infections. Actually, asymptomatic bacteriuria is the most common infection in up to 8% of the population. Symptomatic infection may cause cystitis or include the renal calyces and parenchyma and cause pyelonephritis. There are few common protocols for bacteriuria treatment. The recurrence rate after treatment is 30%. Preventive treatment with nitrofurantoin has been demonstrated to be effective, although there is a small risk to acute respiratory distress which resolved with cessation of the treatment. Renal infection is the most common serious infection during pregnancy. Complication of renal infection can lead to ARDS or urosepsis. Renal infection usually develops during the second trimester and has been related to prim parity and young women.

About 20% of women will deteriorate to renal insufficiency. 30-40% of cases will be followed with recurrent bacteriuria later on, for this reason, a preventive treatment is recommended until delivery. In previous studies the preventive treatment reduced the bacteriuria rate from 38% to 8%.

After delivery, the morphological changes including edema, bladder hyperemia and a raise in the urinary volume, pass away up to 3 months post partum. There is only slight information regarding the rate of bacteriuria during puerperium, most of the information relates to the early puerperium period. In addition, the consequences of such infection are unknown.

The aim of this study is to estimate the efficacy of preventive antibiotic treatment during the puerperium.

Objectives

1. To estimate the rate of bacteriuria and other urinary tract infections during the puerperium among women that had recurrent UTIs or pyelonephritis during pregnancy
2. To evaluate the efficacy of preventive treatment during the puerperium Hypothesis: The pregnancy modifications which cause more urinary tract infections during pregnancy, exist also during the puerperium, and can cause complications Study design Prospective, randomized, open label Study population: Pregnant women with two or more episodes of bacteriuria or one episode of pyelonephritis.

Study period From after delivery to 6 weeks after delivery The study size has been determined according to a reduction in the bacteriuria rate following preventive treatment from 38% to 8%. Basing on that fact, each group has to include 37 women, to get a 80% power with α=0.05.

Study protocol: women will be randomized at recruitment. Demographic and obstetrical data will be collected. The women in the treatment group will receive a prophylactic treatment after delivery for 6 weeks. If the woman breastfeeds, the treatment will be fitted to the situation. Urine culture will be collected in the morning following recruitment, 3 and 6 weeks post delivery. Details regarding bacteriuria, urinary tract infections, pyelonephritis and admissions for related complications will be collected.

The study was approved by the local Helsinki committee.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with two or more episodes of bacteriuria or one episode of pyelonephritis during pregnancy.

Exclusion Criteria:

* Women with malformations of the urinary tract
* women with risk factors to urinary tract infections, for example DIABETES MELLITUS, REFLUX.
* Women with urinary tract infection caused by resistant bacteria (to conventional treatment)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Urinary tract complications | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dep of OG/GYN, Emek Medical Center, Afula, Israel